CLINICAL TRIAL: NCT01580735
Title: A Phase 2, Multicenter, Open-label, Single-arm Study of ARQ 197 Plus Erlotinib in Patient With Locally Advanced or Metastatic EGFR Mutation-positive Non-small-cell Lung Cancer
Brief Title: ARQ 197 Plus Erlotinib in Patient With Locally Advanced or Metastatic EGFR Mutation-positive Non-small-cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 197-007; 23-4882 (Registry Identifier: Pharmaceuticals and Medical Devices Agency)
Record Dates: First submitted 2012-04-16; First posted 2012-04-19 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Non-small-cell Lung Cancer
Keywords: NSCLC; c-MET; EGFR mutation-positive; gefitinib; erlotinib; EGFR-TKI resistance
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARQ 197 (Experimental)
  Interventions: Drug: ARQ 197

INTERVENTIONS:
Drug: ARQ 197 — ARQ 197:360 mg bid (CYP2C19 EM) or 240mg bid (CYP2C19 PM)
  erlotinib: 150 mg qd

SUMMARY:
The primary objective of this study is to examine if the combination regimen of ARQ 197 with erlotinib is active in subjects with locally advanced or metastatic NSCLC with activating mutation EGFR who progressed on EGFR-TKI monotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed surgically unresectable locally advanced or metastatic (stage IIIB/IV) NSCLC with EGFR activating mutation.
* Measurable disease and documented disease progression following the first and immediate EGFR-TKI monotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function

Key Exclusion Criteria:

* Prior therapy with a c-Met inhibitor.
* Any systemic anti-tumor treatment for NSCLC within 7 days prior to randomization.
* Major surgical procedure within 4 weeks prior to randomization
* Known symptomatic brain metastases.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | Up to 6 months
  To examine the objective response rate of ARQ 197 plus erlotinib in advanced/metastatic EGFR-mutated NSCLC, given to patients who previously received erlotinib or gefitinib.

SECONDARY OUTCOMES:
To examine the progression free survival | 30 months
  To examine the progression free survival of patients receiving ARQ 197 plus erlotinib in advanced/metastatic EGFR-mutated NSCLC, given to patients who previously received erlotinib or gefitinib
To examine the overall survival | 30 months
  To examine the overall survival of patients receiving ARQ 197 plus erlotinib in advanced/metastatic EGFR-mutated NSCLC, given to patients who previously received erlotinib or gefitinib
To examine the disease control rate | 30 months
  To examine the disease control rate of patients receiving ARQ 197 plus erlotinib in advanced/metastatic EGFR-mutated NSCLC, given to patients who previously received erlotinib or gefitinib
To estimate the safety profile | 30 months
  To estimate the safety profile of patients receiving ARQ 197 plus erlotinib in advanced/metastatic EGFR-mutated NSCLC, given to patients who previously received erlotinib or gefitinib

CONTACTS AND LOCATIONS:
Locations (1):
- Arakawa-ku, Tokyo, Japan

REFERENCES:
- [Derived] Azuma K, Hirashima T, Yamamoto N, Okamoto I, Takahashi T, Nishio M, Hirata T, Kubota K, Kasahara K, Hida T, Yoshioka H, Nakanishi K, Akinaga S, Nishio K, Mitsudomi T, Nakagawa K. Phase II study of erlotinib plus tivantinib (ARQ 197) in patients with locally advanced or metastatic EGFR mutation-positive non-small-cell lung cancer just after progression on EGFR-TKI, gefitinib or erlotinib. ESMO Open. 2016 Jul 21;1(4):e000063. doi: 10.1136/esmoopen-2016-000063. eCollection 2016. PMID 27843623